CLINICAL TRIAL: NCT06385275
Title: The Role of Vitamin K on Knee Osteoarthritis Outcomes
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-44897; K23AR082938 (NIH)
Record Dates: First submitted 2024-04-21; First posted 2024-04-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Osteo Arthritis Knee
Keywords: Vitamin K-1; Vitamin K-2; Menaquinone-7 (MK-7); Uncarboxylated matrix Gla protein (ucMGP); Phylloquinone
MeSH Terms: interventions — Vitamin K 1; Vitamin K 2; Sugars

STUDY DESIGN:
Intervention Model Description: A stratified permuted block randomization will be used to assign 55 participants in a 1:1:1:1 ratio to each intervention arm. A random allocation sequence will be generated by computer in blocks of 4 or 8, stratified by sex and race.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Use of a placebo from Johnson Compounding Pharmacy (Waltham, MA) of similar appearance and taste to the vitamin K supplements will allow for masking of participants, the study PI, and other study team members to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Vitamin K1 500 µg (Experimental): Participants randomized to this arm will take one Vitamin K1 500 µg pill daily for 4 weeks.
  Interventions: Drug: Vitamin K1 500 µg
- Vitamin K1 1000 µg (Experimental): Participants randomized to this arm will take one Vitamin K1 1000 µg pill daily for 4 weeks.
  Interventions: Drug: K1 1000 µg
- Vitamin K2 (MK-7) 300 µg (Experimental): Participants randomized to this arm will take one Vitamin K2 (MK-7) 300 µg pill daily for 4 weeks.
  Interventions: Drug: Vitamin K2 (MK-7) 300 µg
- Placebo (Placebo Comparator): Participants randomized to this arm will take 1 placebo pill daily for 4 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin K1 500 µg — One pill daily for 4 weeks.
  Other Names: Phylloquinone 500 µg
  Arms: Vitamin K1 500 µg
Drug: K1 1000 µg — One pill daily for 4 weeks.
  Other Names: Phylloquinone 1000 µg
  Arms: Vitamin K1 1000 µg
Drug: Vitamin K2 (MK-7) 300 µg — One pill daily for 4 weeks.
  Other Names: Menaquinone 300 µg
  Arms: Vitamin K2 (MK-7) 300 µg
Other: Placebo — Placebo pill daily for 4 weeks.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The appropriate form and dosing of vitamin K to benefit relevant outcomes in knee osteoarthritis (OA) are not known. In intervention studies for conditions other than knee OA (e.g., prevention of cardiovascular disease), the most commonly used forms and doses include phylloquinone (vitamin K1; 1000µg or 500µg daily) or menaquinone-7 (MK-7 or vitamin K2; 300µg daily). However, whether these doses are adequate to increase vitamin K to levels that ameliorate risk of adverse OA outcomes is not known. Furthermore, although some studies suggest enhanced bioavailability of MK-7 over vitamin K1, as well as extra-hepatic effects, whether this is relevant for an older population with knee OA is not known,

The overall goal of this pilot randomized clinical trial (RCT) is to test different subtypes and doses of vitamin K supplementation in older adults with knee OA and to measure changes in relevant biochemical measures.

ELIGIBILITY:
Inclusion Criteria:

* ≥60 years old
* Clinical diagnosis of knee OA by the treating rheumatologist
* English fluency

Exclusion Criteria:

* Anticoagulation use (including warfarin, dabigatran, rivaroxaban, apixaban)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in uncarboxylated matrix Gla protein (ucMGP) levels | Baseline, 4 weeks
  Plasma ucMGP levels will be measured from blood samples using an enzyme-linked immunoassay (ELISA).
Change in phylloquinone levels | Baseline, 4 weeks
  Plasma phylloquinone will be measured using high-pressure liquid chromatography (HPLC).
Sufficient phylloquinone levels | Baseline, 4 weeks
  Defined as the the proportion of participants achieving phylloquinone level of >1.0 nmol/L, which is the level achieved when adequate intakes are met.
Change in menaquinone-7 (MK-7) levels | Baseline, 4 weeks
  Menaquinone-7 (MK-7) will be measured from blood samples using HPCL.

SECONDARY OUTCOMES:
Study adherence | 4 weeks
  Adherence wil be assessed by analyzing pill counts for each participant.
Participant acceptability of intervention | 4 weeks
  Participants will use a 5 point LIkert scale to rate acceptability of the overall study, the pill tste, gastrointestinal tolerance, burden, and blood collection.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Liew, MD MS, Principal Investigator — Boston University Chobanian & Avedisian School of Medicine, Department of Rheumatology
Locations (1):
- Boston Medical Center, Rheumatology Clinic, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No